CLINICAL TRIAL: NCT03051360
Title: Proprotein Convertase Subtilisin Kexin Type 9 Inhibitor in Aortic Stenosis
Brief Title: PCSK9 Inhibitors in the Progression of Aortic Stenosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Soo Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PCSK9 AS
Record Dates: First submitted 2017-01-23; First posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Aortic Valve Stenosis
Keywords: aortic valve stenosis; PCSK9 inhibitor
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — erucylphosphocholine

STUDY DESIGN:
Intervention Model Description: Prospective, Double blind, Multi-center, Randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PCSK9 inhibitor (Active Comparator): Patients will receive bi-weekly PCSK9 inhibitor .
  Interventions: Drug: PCSK9 Inhibitor [EPC]
- Placebo (Placebo Comparator): Patients will receive bi-weekly placebo.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: PCSK9 Inhibitor [EPC] — Patients will receive PCSK9 inhibitor by a biweekly injection
  Arms: PCSK9 inhibitor
Drug: Placebos — Patients will receive Placebo by a biweekly injection
  Arms: Placebo

SUMMARY:
Investigators plan evaluate whether PCSK9 inhibitors, a medication that can lower lipoprotein(a) and control dyslipidemia, can inhibit the progression of aortic stenosis, through a randomized controlled trial.

DETAILED DESCRIPTION:
Aortic valve disease is the most common form of heart valve disease and is a major burden to society. Aortic valve disease is also expected to become more prevalent with the aging. Among aortic diseases, 'aortic stenosis (AS)', which is a narrowing of the aortic valve, and leads to symptoms of heart failure and sometimes death.

For treatment of AS, the valve in replaced in a surgical to percutaneous method. Regardless of the method, valve replacement has its potential costs and complications that is an important issue that needs to be solved. Therefore, controlling the progression of AS and increasing the efficacy of medical therapy before valvular replacement is needed, is an important medico-social problem.

Regarding the pathophysiology of AS, an elevation of lipoprotein(a) and dyslipidemia have been reported to be associated with the progression of cardiovascular calcification.

PCSK9 inhibitors, which is a medication that can control both lipoprotein(a) and dyslipidemia may be a effective medication to control the progression of AS.

Therefore, investigators will perform a randomized control trial, to compare the effect of PCSK9 inhibitors vs. placebo in its influence to AS progression.

ELIGIBILITY:
Inclusion Criteria:

1. The patient agrees to participate in this study by signing the informed consent form. Alternatively, a legally authorized patient representative may agree to the patient's participation in this study and sign the informed consent form.
2. The patient has a working diagnosis of aortic stenosis (mild to moderate), and has fair treatment compliance.

Exclusion Criteria:

1. Age under 19 years old
2. Hypersensitivity to PCSK9 inhibitor
3. LDL cholesterol < 70mg/dL at baseline
4. Poor treatement compliance (The patient will need to visit the out-patient clinic every 2-weeks for medication)
5. Positive pregnancy test or is known to be pregnant
6. Any other reason the investigator deems the subject to be unsuitable for the study (e.g., Active malignant tumor, Any life-threatening condition with life expectancy less than 6months, etc.)
7. Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the investigator, would preclude safe completion of the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression of the Calcium score measured by cardiac CT (Agatston score) and by NaF PET | 2 years
  Calcium score progression in the PCSK9 inhibitor group and placebo group

SECONDARY OUTCOMES:
Efficacy of inhibition in calcium score progression (Agatston score) by the presence of Lp(a) SNPs | 2 years
Mean change in Lp(a) levels between treatment arms | 2 years
  Lp(a) levels will be measured in blood chemistry
Mean change in lipid panel (LDL, HDL, TG, Cholesterol) level | 2 years
  Lipid panels will be measured in blood chemistry
Aortic valve area measured by echocardiography | 2 years
Aortic valve peak velocity measured by echocardiography | 2 years
Any death event | 2 years
Any cardiac death event | 2 years
Any myocardial infarction event | 2 years
Any revascularization for coronary artery disease | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided